CLINICAL TRIAL: NCT02778451
Title: Certification Standards and Diagnostic Accuracy for Surgeon-performed Ultrasonography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Tobias Todsen, M.D., Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-3-2013-081
Record Dates: First submitted 2016-04-08; First posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Ultrasonography Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasonography-experienced surgeons (Other): Attending physicians and consultants in head and neck surgery using head and neck Ultrasonography on a daily basis.
  Interventions: Other: Measurement of competence
- Ultrasonography novices (Other): Physicians participating in their one-year internship at other surgical or medical departments with no experience with head and neck US or head and neck surgery.
  Interventions: Other: Measurement of competence

INTERVENTIONS:
Other: Measurement of competence — This study is a psychometric validation of a generic assessment tool to evaluate ultrasonography competence among surgeons

SUMMARY:
Ultrasonography (US) is an operator depended image modality that is difficult to reproduce and interpret by others. Competence of the US operator is crucial for reliable diagnostics but no evidence-based certification of head and neck US skills has been developed. Investigators conducted an experimental study aimed to explore diagnostic accuracy and establish validity evidence for certification standards in surgeon-performed ultrasonography.

ELIGIBILITY:
1. Ultrasonography-experienced surgeons

   Inclusion Criteria:
   * Board certified otolaryngologist
   * Daily use of head and neck Ultrasonography
2. Ultrasonography novices:

Inclusion Criteria:

* Medical doctor during internship

Exclusion Criteria:

* experience with head and neck Ultrasonography
* experience with head and neck surgery

Ages: 26 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Competence score on a generic skills assessment scale (The Objective Structured Assessment of Ultrasound Skills (OSAUS)) | up to 24 months
  Performance were video-recorded Maj 25, 2013 and afterwards assessed by a consultant in diagnostic radiology and a consultant in head and neck surgery

SECONDARY OUTCOMES:
Diagnostic accuracy assessed by a head and neck surgeon reading the ultrasonography report | up to 24 months
  Assessed by a head and neck surgeon reading the ultrasonography report of the participating physicians from the experimental study conducted Maj 25, 2013

IPD SHARING:
Plan to Share IPD: No